CLINICAL TRIAL: NCT04711434
Title: PD-1 Antibody for the Prevention of Adenomatous Polyps and Second Primary Tumors in Patients With Lynch Syndrome: An Open-label, Multicenter, Randomized Controlled Clinical Trial
Brief Title: PD-1 Antibody for The Prevention of Adenomatous Polyps and Second Primary Tumors in Lynch Syndrome Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Fujian Cancer Hospital (Other Government); Guangdong Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); The Third Affiliated Hospital of Kunming Medical College. (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2020-059-01
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Lynch Syndrome
Keywords: Toripalimab; Lynch Syndrome; Prevention
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — spartalizumab; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention group (Experimental): Toripalimab: 240mg IV every 3 months for a year
  Interventions: Drug: PD-1 Antibody
- Follow-up group (No Intervention): Routine follow-up, no intervention

INTERVENTIONS:
Drug: PD-1 Antibody — Toripalimab: 240mg IV every 3 months for a year
  Other Names: Toripalimab
  Arms: Prevention group

SUMMARY:
This study aims to explore the role of PD-1 Antibody in preventing adenomatous polyps and second primary tumors in patients with Lynch Syndrome. There two arms, one is the experimental arm (PD-1 antibody prevention group) and the other is the control arm (routine follow-up group). For the experimental group, Tripleitriumab (PD-1 antibody) is given every 3 months for a year.

DETAILED DESCRIPTION:
Lynch syndrome (LS) is a hereditary cancer syndrome that causes the majority of hereditary CRC and approximately 3% of all CRC. LS significantly increases the risk for an individual to develop CRC during their lifetime. Individuals with LS also have an increased risk to develop extracolonic cancers, including endometrial, gastric, ovarian, upper urinary tract, small bowel, biliary tract, CNS, and certain types of skin cancer. Given the hereditary nature of this syndrome, preventing second primary tumors in patients with Lynch Syndrome after surgery to the primary site is very important.

The purpose of this study is to prevent adenomatous polyps and second primary tumors using PD-1 antibody (Tripleitriumab) in patients with Lynch Syndrome.

The primary outcome of this study is the incidence of intestinal adenomatous polyps and secondary primary tumors. The secondary outcomes are the incidence of colorectal adenomatous polyps greater than 1cm, incidence of high-grade colorectal polyps, treatment-related adverse events, disease-free Survival and overall Survival.

There are two groups: the PD-1 antibody prevention group and the routine follow-up group. For the PD-1 antibody prevention group, participants will receive Toripalimab 240mg IV every 3 months for a year. For the routine follow-up group, there is no drug intervention.

This whole study will take 5 years: the first year for recruiting and the latter four years for follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Lynch syndrome with germline variants of MLH1, MSH2, or EPCAM (pathogenic or likely pathogenic variants)
2. Necessary treatments have been done, such as surgery, chemotherapy, radiation therapy, etc.
3. Have a resection, including right hemicolectomy, left hemicolectomy, sigmoid colectomy, or anterior resection of rectal cancer, or endoscopic adenoma resection
4. Aged 18-70 years old
5. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
6. White blood cell (WBC) > 4000/mm3, Platelet count >100000/mm3, HB >10 g/dL
7. Serum glutamic-oxaloacetic transaminase (SGOT) < 1.5 × the upper limit of normal (ULN), Serum glutamic pyruvic transaminase (SGPT) < 1.5 × ULN prior to randomization, Total bilirubin (TBIL) < 1.5 mg/dL
8. Serum creatinine (Scr) <1.8 mg/dL

Exclusion Criteria:

1. Lynch syndrome with germline variants of MSH6 and PMS2
2. Previous immunotherapy has been taken, such as anti-PD-1, anti-PD-L1, etc.
3. Long-term use of aspirin
4. Suffering from autoimmune diseases
5. Active infection with hepatitis B or hepatitis C (high copy number of viral DNA) or human immunodeficiency virus (HIV)
6. Other clinically serious active infections (NCI-CTC 4.0)
7. With cachexia or organ dysfunction
8. Suffering from seizures requiring treatment (such as steroids or antiepileptic therapy)
9. Unable to participate or complete the study due to substance abuse, or medical, psychological, or social disorder
10. Known allergy to any drugs in this study
11. Pregnant or nursing women, or women of childbearing potential who are not using adequate contraception
12. Any unstable condition or situation that could compromise the safety and compliance of participants.
13. Failure to sign an informed consent form

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients from randomization to the first appearance of one of the following: adenomatous polyps or second primary tumors | up to 5 years

SECONDARY OUTCOMES:
The percentage of patients developing polyps greater than 1cm within 5 years from randomization | up to 5 years
The percentage of patients developing high-grade polyps on pathology within 5 years from randomization. | up to 5 years
Treatment-related adverse events | up to 5 years
  Incidence and severity of adverse events as assessed by NCI CTCAE V4.0
Effectiveness with different genotypes or phenotypes | up to 5 years
  Estimated the percentage of patients with different genotypes or phenotypes not developing polyps or second primary tumors within 5 years from randomization.
Disease-free Survival | up to 5 years
  defined as the time from randomization to the first appearance of one of the following: primary tumor recurrence, or death without cancer event; or censored at date of last follow-up
Overall Survival | up to 5 years
  defined as the time from randomization to death from any cause. Participants who were alive or lost to follow-up at the time of the analysis were censored at the date they were last known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Peirong Ding, MD, Ph D, Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong, China